CLINICAL TRIAL: NCT00877903
Title: A Phase II, Multi-center, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of PROCHYMAL® (Ex Vivo Cultured Adult Human Mesenchymal Stem Cells) Intravenous Infusion Following Acute Myocardial Infarction
Brief Title: Prochymal® (Human Adult Stem Cells) Intravenous Infusion Following Acute Myocardial Infarction (AMI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mesoblast, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mesoblast, Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 403
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Myocardial Infarction
Keywords: Acute myocardial infarction; AMI; Myocardial infarction; Heart attack; Mesenchymal stem cells; MSC; Adult human stem cells; Osiris
MeSH Terms: conditions — Myocardial Infarction | interventions — remestemcel-l

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Prochymal® (Experimental): Participants will receive Prochymal® single intravenous (IV) infusion at a dose of 200 x 10^6 human mesenchymal stem cells (hMSC), reconstituted in 80 mL, delivered at a rate of 2 mL/min, with a maximum rate of 5.0 x 10^6 hMSC/minute, and the participants will be followed for 24 months and remain in the study for up to 60 months.
  Interventions: Drug: Prochymal®
- Placebo (Placebo Comparator): Participants will receive Prochymal® placebo-matching single IV infusion at a dose of of 200 x 10^6 hMSC, reconstituted in 80 mL, delivered at a rate of 2 mL/min, with a maximum rate of 5.0 x 10^6 hMSC/minute, and the participants will be followed for 24 months and remain in the study for up to 60 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prochymal® — Intravenous infusion of ex vivo cultured adult human mesenchymal stem cells
  Other Names: Remestemcel-L
  Arms: Prochymal®
Drug: Placebo — Intravenous infusion of excipients of Prochymal®
  Arms: Placebo

SUMMARY:
The objective of the present study is to establish the safety and efficacy of Prochymal® following first acute myocardial infarction.

DETAILED DESCRIPTION:
The standard of care treatment for acute myocardial infarction (AMI) usually includes immediate perfusion, optimal pain relief, oxygen, aspirin or other anti-coagulants, Beta-Blockers, nitrates and Ace-inhibitors. However, because salvaging the viable myocardium is dependent on early reperfusion, only a minority of participants will reach the hospital within the time-window for myocardial rescue. Thus, even if the participant manages their tobacco use, hypertension, lipid levels, diabetes, weight and exercise, many participants will go on to develop Congestive Heart Failure (CHF). Though the medical management for CHF may improve symptoms and slow disease progression, such treatment cannot restore a functioning myocardium. A therapy that could improve the myocardial remodeling process and reduce the incidence or severity of CHF following acute MI would provide a significant benefit. The characteristics and biologic activity of Prochymal®, along with a good safety profile in human trials to date, suggest that Prochymal® may be a good candidate for addressing this unmet medical need.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 21 and 85 years old, inclusive
* First heart attack within 7 days prior to randomization and drug infusion
* Baseline left ventricular ejection fraction (LVEF) 20-45%
* Hemodynamically stable within 24 hours prior to randomization
* Adequate pulmonary function

Exclusion Criteria:

* Previous medical history of heart attack, heart failure, significant valvular heart disease, aortic dissection
* Pacemaker or other device
* Pregnant, breast-feeding, or intends to become pregnant during the study
* Allergy to cow or pig derived products
* Evidence of active malignancy or prior history of active malignancy
* Major surgical procedure or major trauma within the past 14 days
* Autoimmune disease (e.g., Lupus, Multiple Sclerosis)
* Any medical condition, which in the opinion of the Investigator, renders participation unsuitable
* Undergone pharmacologic cardioversion or external defibrillation within 24 hours of randomization.
* Experienced cardiac arrest more than 36 hours after presentation to site or within 24 hours of randomization.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2009-03-30 (Actual); Primary Completion 2011-05-18 (Actual); Study Completion 2016-03-14 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Cardiac Magnetic Resonance (CMR) imaging-determined End Systolic Volume (ESV) at Month 3 | Baseline, Month 3

SECONDARY OUTCOMES:
Left Ventricular End Systolic Volume | 6 months
Infarct Size | 3 and 6 months
Left Ventricular Ejection Fraction | 3 and 6 months
Left Ventricular End Diastolic Volume | 3 and 6 months
Number of Participants with Ventricular Arrhythmias | 3 and 6 months
Duke Activity Status Index (DASI) Assessment | 6, 12, and 24 months
  The Duke Activity Status Index (DASI) is a brief, self-administered questionnaire that provides a standardized assessment of functional status and quality-of-life that correlates well with an objective measure of maximal exercise capacity. The scale ranges from 0 (unable to perform any tasks) to 58.20 (able to perform all tasks). Higher scores indicate a greater ability to perform daily activities.
New York Heart Association (NYHA) Congestive Heart Failure Classification Status | 6, 12, 24, and 60 months
Maximal Symptom-limited Exercise Test (Treadmill) | 6 and 12 months
Number of Participants with Major Adverse Cardiac Events (MACE) | 6, 12, 24, and 60 months
Overall Survival | 60 months
Number of Participants with Adverse Events | 3,6,12,24,60 months

CONTACTS AND LOCATIONS:
Overall Officials: Ken Borow, MD, Study Director — Mesoblast, Inc.
Locations (33):
- United States (32):
  - Mercy Gilbert Medical Center / Catholic Health Care West, Gilbert, Arizona
  - University of Arizona, Tucson, Arizona
  - UC Davis Medical Center, Sacramento, California
  - University of California - San Diego (UCSD), San Diego, California
  - University of Miami, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Rush University Medical Center, Chicago, Illinois
  - The Care Group, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Cotton-O'Neil Clinical Research Center, Topeka, Kansas
  - University of Maryland Hospital, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
  - Michigan Cardiovascular Institute, Saginaw, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - University at Buffalo - Buffalo General Hospital, Buffalo, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - The Lindner Research Center, Cincinnati, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Penn State University - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - The Stern Cardiovascular Center, Germantown, Tennessee
  - Austin Heart P.A., Austin, Texas
  - University of Texas Health Science Center, Houston, Texas
  - Fletcher Allen Health Care, Burlington, Vermont
  - University of Wisconsin School of Medicine, Madison, Wisconsin
- McGill University Health Centre, Montreal, Quebec, Canada